CLINICAL TRIAL: NCT03764865
Title: Day 3 vs Day 5 Embryo Transfer for Patients With Low Embryo Numbers Going Through in Vitro Fertilization (PILOT STUDY)
Brief Title: PooR Embryo Yield Cleavage Stage Versus blaStocyst Embryo Transfer (PILOT STUDY)
Acronym: PRECiSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston IVF (Other)
Responsible Party: Principal Investigator, Werner Neuhausser, Instructor in Obstetrics, Gynecology and Reproductive Biology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000530
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Infertility
Keywords: cleavage embryo; blastocyst; embryo transfer; in vitro fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: non-inferiority
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- day 3 embryo transfer (Experimental): embryo transfer 3 days after fertilization
  Interventions: Procedure: day 3 uterine transfer
- day 5 embryo transfer (Experimental): embryo transfer 5 days after fertilization
  Interventions: Procedure: day 5 uterine transfer

INTERVENTIONS:
Procedure: day 3 uterine transfer — uterine transfer of embryo on day 3 after fertilization (cleavage stage)
  Arms: day 3 embryo transfer
Procedure: day 5 uterine transfer — uterine transfer of embryo on day 5 after fertilization (blastocyst stage)
  Arms: day 5 embryo transfer

SUMMARY:
The purpose of this small-scale pilot study (10 patients) is to test the study protocol for an RCT comparing IVF outcomes between day 3 and day 5 embryo transfer in patients with five or fewer embryos in a fresh embryo transfer in vitro fertilization (IVF) cycle. Information derived from this RCT would allow us to maximize the chances of success for these patients undergoing IVF.

DETAILED DESCRIPTION:
Embryos created with assisted reproductive technology (ART, e.g. in vitro fertilization (IVF)) are commonly transferred into a woman's uterus at either the cleavage stage (day 3 after egg retrieval) or blastocyst stage (day 5 after egg retrieval). Until recently, most IVF cycles transferred embryos at the cleavage stage. However, with improvements in in vitro culture technique there has been a steady shift in practice to transfer embryos at the blastocyst stage (day 5 after egg retrieval) as this timing is about the same as when embryos reach the endometrial cavity in natural conception.

There now is a general consensus that, for good prognosis patients, those with a high embryo from the IVF cycle, it is beneficial to transfer the embryo on day 5 rather than day 3. The rationale for this is to allow for self-selection of embryos, meaning those that develop to blastocyst in vitro are more likely to be viable in vivo and result in a viable pregnancy. In addition, transferring an embryo on day 5 improves uterine/embryonic synchronicity and thereby improves outcomes. This allows the transfer of fewer embryos and decreases the likelihood of multiples (twins, triplets, etc.).

As a result, day 5 transfer has become standard of care for good prognosis patients in the United States. The American Society of Reproductive Medicine1 issued a committee opinion in 2013 to this effect stating that in "good prognosis" patients, blastocyst transfer results in a significant increase in live birth rates compared to transfer of an equal number of cleavage stage embryos (50.5% vs. 30.1%, P< .01)2-5. In addition, for unselected and poor prognosis patients, no high-quality studies have evaluated whether blastocyst transfer increases live birth rates when compared to cleavage stage transfer.

It is possible that the attrition of day 3 embryos in vivo is lower than the attrition in vitro and that day 5 transfer leads to loss of embryos that may have survived in vivo. In addition, women undergoing blastocyst culture are expected to have a higher incidence of cycle cancellation due to failure of the embryo to develop to a blastocyst6 and of having fewer embryos cryopreserved (frozen)7. Because of this, in Europe and Asia, day 3 transfer is the most common practice.

On the other hand, transferring embryos on day 3 decreases our ability to select the best embryo, increases laboratory costs and may increase multiple pregnancy rates as, typically, more embryos are transferred at this time. In addition, in vivo, day 3 embryos are in transit through the fallopian tube during natural conception and are exposed to a different developmental and nutritional environment than day 3 IVF embryos transferred into the uterine cavity. Thus, it is possible that exposing day 3 embryos to the physiologically premature uterine environment (particularly one that has been subjected to superovulation and thus high levels of estrogen) increases embryo attrition compared to day 5 transfer, particularly in poor prognosis patients.

Therefore, a clinical dilemma exists for poor prognosis patients (those with ≤5 embryos available on day 1 after egg retrieval). Currently, many practices in the United States transfer embryos from these patients on day 3 due to the risk of not having embryos available to transfer on day 5. Any remaining embryos are then frozen if they meet criteria on day 5/6.

Retrospective data from Boston IVF, BIDMC's affiliated infertility treatment center, demonstrates that the live birth rate per transfer among poor prognosis patients is 18% among those who have a cleavage stage transfer and 38% among those who have a blastocyst transfer.

At Boston IVF, about 35% of patients have a day 3 embryo transfer, which is consistent with national trends. For a patient undergoing an IVF cycle at Boston IVF, a physician may choose to transfer an embryo on day 3 or day 5 or allow the laboratory to make that decision, based on the number of embryos the patient has on day 1 after egg retrieval and the patient's age. This decision typically is made prior to the IVF cycle. As demonstrated above, pregnancy rates are far lower in the cleavage stage transfer group and there is the possibility that, within a select cohort of these patients, we are unrealistically raising patient's expectations of a live birth.

The purpose of this study is to compare IVF outcomes among poor prognosis patients (≤5 embryos with two pronuclei) who have a day 3 transfer to those who have a day 5 transfer.

ELIGIBILITY:
Inclusion Criteria:

* First autologous IVF cycle
* Written, informed consent

Exclusion Criteria:

* Planned gestational carrier
* Planned donor egg
* Morbid obesity: BMI >40
* History of recurrent pregnancy loss (≥2 spontaneous abortions)
* Presence of uterine factor infertility
* Treatment plan includes embryos cultured 'out of protocol'
* Planned preimplantation genetic testing

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
live birth | 9 months
  defined as delivery of a live born infant ≥22 weeks of gestation

SECONDARY OUTCOMES:
Clinical pregnancy | 14 days
  defined by confirmation of a gestational sac on ultrasound
Ongoing pregnancy | 9 months
  defined by ultrasound confirmation of a gestational sac with at least one fetal pole with a fetal heartbeat
Multiple pregnancy | 9 months
  defined as twins or higher-order gestations
Time to pregnancy/live birth | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Werner Neuhausser, MD PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Practice Committees of the American Society for Reproductive Medicine and the Society for Assisted Reproductive Technology. Blastocyst culture and transfer in clinical-assisted reproduction: a committee opinion. Fertil Steril. 2013 Mar 1;99(3):667-72. doi: 10.1016/j.fertnstert.2013.01.087. PMID 23714439
- [Background] Gardner DK, Schoolcraft WB, Wagley L, Schlenker T, Stevens J, Hesla J. A prospective randomized trial of blastocyst culture and transfer in in-vitro fertilization. Hum Reprod. 1998 Dec;13(12):3434-40. doi: 10.1093/humrep/13.12.3434. PMID 9886530
- [Background] Glujovsky D, Farquhar C, Quinteiro Retamar AM, Alvarez Sedo CR, Blake D. Cleavage stage versus blastocyst stage embryo transfer in assisted reproductive technology. Cochrane Database Syst Rev. 2016 Jun 30;(6):CD002118. doi: 10.1002/14651858.CD002118.pub5. PMID 27357126
- [Background] Papanikolaou EG, D'haeseleer E, Verheyen G, Van de Velde H, Camus M, Van Steirteghem A, Devroey P, Tournaye H. Live birth rate is significantly higher after blastocyst transfer than after cleavage-stage embryo transfer when at least four embryos are available on day 3 of embryo culture. A randomized prospective study. Hum Reprod. 2005 Nov;20(11):3198-203. doi: 10.1093/humrep/dei217. Epub 2005 Jul 29. PMID 16055454
- [Background] Papanikolaou EG, Camus M, Kolibianakis EM, Van Landuyt L, Van Steirteghem A, Devroey P. In vitro fertilization with single blastocyst-stage versus single cleavage-stage embryos. N Engl J Med. 2006 Mar 16;354(11):1139-46. doi: 10.1056/NEJMoa053524. PMID 16540614
- [Background] Marek D, Langley M, Gardner DK, Confer N, Doody KM, Doody KJ. Introduction of blastocyst culture and transfer for all patients in an in vitro fertilization program. Fertil Steril. 1999 Dec;72(6):1035-40. doi: 10.1016/s0015-0282(99)00409-4. PMID 10593377
- [Background] Tsirigotis M. Blastocyst stage transfer: pitfalls and benefits. Too soon to abandon current practice? Hum Reprod. 1998 Dec;13(12):3285-9. doi: 10.1093/humrep/13.12.3285. No abstract available. PMID 9886498
- [Derived] Neuhausser WM, Vaughan DA, Sakkas D, Hacker MR, Toth T, Penzias A. Non-inferiority of cleavage-stage versus blastocyst-stage embryo transfer in poor prognosis IVF patients (PRECiSE trial): study protocol for a randomized controlled trial. Reprod Health. 2020 Jan 30;17(1):16. doi: 10.1186/s12978-020-0870-y. PMID 32000803